CLINICAL TRIAL: NCT07000864
Title: Predicting Response to Therapy From Analysis of Live Tumor Fragments of Surgical Resections
Brief Title: A Study of Live Tumor Fragments of Surgical Resections
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Debabrata Mukhopadhyay, PhD, Principal Investigator, Mayo Clinic
Other Study IDs: MC250101; 25-002240 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2025-05-23; First posted 2025-06-03 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Cancer; Tumor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: No intervention — Lab-based correlative study; no intervention

SUMMARY:
The purpose of this study is to obtain unused resected tumor tissue sample and associated clinical data from patients enrolled in this study to research ex vivo treatment response and integrity of tumor microenvironment using omics analysis and imaging while maintaining cell stability in a live environment.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and sign informed consent
* Planning to undergo a surgical procedure to remove cancer

Exclusion Criteria:

* Does not meet Inclusion criteria
* No tissue for research available at time of surgery

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Male and female patients planning to undergo surgery for removal of cancer at Mayo Clinic in Florida.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Tissue response to treatment | Up to 72 hours
  Tumor sample fragments will be treated with various combination of chemotherapy and immunotherapy drugs that are commonly used to treat patients clinically (panel of drugs will be selected based on cancer type). response to the treatment will be assessed at multiple timepoints during a 72-hour period.

CONTACTS AND LOCATIONS:
Overall Officials: Debabrata Mukhopadhyay, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials